CLINICAL TRIAL: NCT06193070
Title: Escape Room: A Gamified Approach to Learning About Cancer Nutrition Information
Brief Title: An Escape Room Intervention to Help Improve Breast Cancer Patients' Ability to Navigate Online Access to Nutrition Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Megan Shen, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1123830; NCI-2023-08424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20282 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Early Intervention, Educational; Interviews as Topic; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (escape room game) (Experimental): Patients play the virtual misinformation escape room game consisting of 5 puzzles and a final task over 30-45 minutes on study.
  Interventions: Other: Educational Intervention; Other: Interview; Other: Survey Administration; Other: Telemedicine

INTERVENTIONS:
Other: Educational Intervention — Play virtual misinformation escape room game
  Other Names: Escape room cancer nutrition game
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Telemedicine — Play virtual misinformation escape room game
  Other Names: Telehealth

SUMMARY:
This clinical trial evaluates an educational escape room intervention for improving awareness of and concern about breast cancer misinformation and reducing vulnerability to believing cancer misinformation among patients with stage I-III breast cancer. Misinformation, or communication about health information that is inaccurate or false, can have serious health consequences for those that believe it. The rise of the access to and use of various sources of information on the internet such as websites and social media has caused the spread of misinformation and disinformation to grow rapidly, resulting in negative consequences on health outcomes. Cancer misinformation, in particular, has become an increasingly prevalent issue that poses a real threat to the many cancer patients in the United States. The educational escape room intervention is a game designed to teach participants how to discern whether cancer nutrition information is accurate or may potentially be misinformation. Participants are immersed in the narrative while solving puzzles to learn key themes such as the need to talk to their doctors, looking for scientific studies, as well as avoiding fads and trends, miracle cures, anecdotal evidence, and targeted and clickbait ads.

DETAILED DESCRIPTION:
OUTLINE:

Patients complete a baseline before playing the virtual cancer nutrition information escape room game. Patients then play the virtual misinformation escape room game consisting of 5 puzzles and a final task over 30-45 minutes on study. Following the escape room game, patients complete a post-game survey and debrief interview (15 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* English speaking
* Able to provide informed consent
* Have access to a computer (desktop or laptop)
* Have been previously diagnosed with breast cancer (Stages I-III) and currently in active treatment for breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Shen, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Escape Room Game: Patients play the virtual misinformation escape room game consisting of 5 puzzles and a post-game debrief over 30-45 minutes on study.
  Educational Intervention: Play virtual misinformation escape room game
  Interview: Ancillary studies
  Survey Administration: Ancillary studies
  Telemedicine: Play virtual misinformation escape room game
Period: Overall Study
Arm/Group | Escape Room Game
Started | 45
Completed | 43
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Total number of participants enrolled who completed baseline.
Groups:
- Escape Room Game: Patients play the virtual misinformation escape room game consisting of 5 puzzles and a final task over 30-45 minutes on study.
  Educational Intervention: Play virtual misinformation escape room game
  Interview: Ancillary studies
  Survey Administration: Ancillary studies
  Telemedicine: Play virtual misinformation escape room game
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Of the n=43 patients who entered baseline data, n=2 entered the date of the survey in the date of birth field, causing missing data on this variable.
  years
    number analyzed (Participants) | 41
    (all) | 52.2 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Accrued to the Study (Feasibility)
Description: The percentage of patients who accrue to the study among those who are eligible and approached.
Time Frame: At enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Escape Room Game
Number analyzed (Participants) | 45
Participants | 45

2. Primary Outcome: Percentage of Patients Who Complete Game Sessions (Feasibility)
Description: The percentage of patients who complete the game.
Time Frame: Up to 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
Participants | 43

3. Primary Outcome: Satisfaction (Acceptability)
Description: Will be assessed using a Likert-type question to assess satisfaction with the game (1 = not at all satisfied, 10 = very satisfied)
Time Frame: Up to 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
units on a scale | 6.8 (2.34)

4. Primary Outcome: Likelihood to Recommend the Game to Someone Else (Acceptability)
Description: Will be assessed using a Likert-type question to assess likelihood to recommend the game to someone else (1 = not at all likely, 5 = very likely).
Time Frame: Up to 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
units on a scale | 3.1 (1.31)

5. Primary Outcome: Usability (System Usability Scale)
Description: Usability will be assessed using the System Usability Scale (SUS). The SUS is a reliable, 10-item measure 10-item scale, scored on a 5-point Likert scale (1=strongly disagree; 5=strongly agree), with previously reported excellent internal reliability (Cronbach's α = 0.91). Total scores on the SUS range from 0-100, with higher scores indicating greater usability.
Time Frame: Up to 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
score on a scale | 59.3 (19.70)

6. Secondary Outcome: Types of Online Information
Description: Will be assessed using a 6-item checklist that asks which resources participants or their family members have used to find nutrition information in the past 3 months (self-care/health and wellness book, telephone advice service, booklet/flyer shared by a health professional, internet forums, internet search, social media).
  Reported as count data of number of participants who endorsed one or more sources (self-care/health and wellness book, telephone advice service, booklet/flyer shared by a health professional, internet forums, internet search, social media).
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
Participants
  Self-care/Health and wellness book | 16
  Telephone advice service | 1
  Booklet/flyer shared by a health professional | 5
  Internet forums | 7
  Internet search | 30
  Social media | 14
  None of the above | 6

7. Secondary Outcome: Concern About Misinformation and Confidence in Identifying Misinformation
Description: Will be assessed using our 4-item scale in which patients indicate degree to which they agree with statements using a 5-point Likert scale (1=strongly disagree, 5=strongly agree). Items asked participants to rate the degree to which they agree with the following: (1) I am more worried about accidentally believing misinformation, (2) I am more worried about accidentally sharing misinformation online, (3) I am more concerned about misinformation in society, and (4) I feel more confident in my ability to identify misinformation).
Time Frame: Up to 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
units on a scale
  (1) I am more worried about accidentally believing misinformation. | 2.1 (1.13)
  (2) I am more worried about accidentally sharing misinformation online. | 2.0 (1.18)
  (3) I am more concerned about misinformation in society. | 3.7 (1.24)
  (4) I feel more confident in my ability to identify misinformation. | 3.6 (0.98)

8. Secondary Outcome: Cancer Nutrition Information Beliefs
Description: Will be assessed using a 15-item checklist of common cancer nutrition misinformation and credible nutrition advice, using a 5-point Likert Scale (1=definitely false, 5 = definitely true). Data reported as an average score at both pre-intervention (pre-game score) and post-intervention (post-game score).
Time Frame: At baseline and up to 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escape Room Game
Number analyzed (Participants) | 43
score on a scale
  Pre-game score | 3.6 (0.68)
  Post-game score | 3.8 (0.73)
Statistical Analysis 1: Comparison: Escape Room Game; All participants were exposed to the intervention, and pre- and post-game scores within subject were examined; Test type: Other — A one-tailed paired t-test was run to examine within subject mean difference on the cancer nutrition information beliefs scale pre- and post-game; p < .001, t-test, 1 sided — The threshold was set at alpha < 0.05; A paired samples t-test was run on pre- and post-game mean scores within subjects

ADVERSE EVENTS:
Time Frame: Each enrolled participant was followed for adverse events at the point of consent until the completion of the final survey, up to 44 days.
Arm/Group | Escape Room Game
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT06193070/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT06193070/ICF_000.pdf